CLINICAL TRIAL: NCT00847678
Title: A Multicenter, Randomized Study to Assess the Efficacy and Safety of Mycograb® as Adjunctive Therapy for Cryptococcal Meningitis in Patients With AIDS
Brief Title: Efficacy and Safety of Mycograb as Adjunctive Therapy for Cryptococcal Meningitis in Patients With AIDS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MYC123A2201; NTP/Mycograb/003B
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Cryptococcal Meningitis
Keywords: Cryptococcal Meningitis
MeSH Terms: conditions — Meningitis, Cryptococcal | interventions — efungumab; Amphotericin B; Flucytosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- 1 (Experimental): Mycograb + Amphotericin B + 5 flucytosine
  Interventions: Biological: Efungumab (Mycograb); Biological: Amphotericin B; Biological: 5 flucytosine
- 2 (Placebo Comparator): Placebo + Amphotericin B + 5 flucytosine
  Interventions: Biological: placebo; Biological: Amphotericin B; Biological: 5 flucytosine
- 3 (Experimental): Mycograb + Amphotericin B
  Interventions: Biological: Efungumab (Mycograb); Biological: Amphotericin B

INTERVENTIONS:
Biological: Efungumab (Mycograb)
  Arms: 1; 3
Biological: placebo
  Arms: 2
Biological: Amphotericin B
Biological: 5 flucytosine
  Arms: 1; 2

SUMMARY:
This is a multicenter, randomized, efficacy and safety trial to evaluate Mycograb®. Subjects will be randomized to one of the 3 arms: 1/ Amphotericin B (0.7 mg/kg/d) plus 5-flucytosine (100 mg /kg/d); 2/ Amphotericin B plus Mycograb® (dosed 1 mg/kg via a central line or peripheral venous line twice daily for 7 consecutive days); 3/ Amphotericin B plus 5-flucytosine plus Mycograb® (dosed 1 mg/kg via a central line or peripheral venous line twice daily for 7 consecutive days). After 2 weeks, all patients will be switched to fluconazole at 400 mg/d for 8 weeks and 200 mg/d thereafter. The total duration of the study will be approximately 24 months

ELIGIBILITY:
Inclusion criteria:

* Male or non-pregnant female who is > 18 years old.
* HIV-positive or unknown, with acute, either first or recurrent episode of cryptococcal meningitis.
* Currently on no treatment, or receiving treatment (< 3 days) with either amphotericin B plus 5-flucytosine, or amphotericin B alone.
* Positive CSF culture for Cryptococcus neoforman.
* Physical signs and symptoms of meningitis, evidenced by one or more of the following: fever, headache, meningeal signs and neurologic findings.

Exclusion criteria:

* Excluded for coma, or significant other medical conditions.
* Subject has other opportunistic fungal infections that requires other systemic antifungal therapies.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-08; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
proportion of patients (receiving Mycograb + Amphotericin B + 5-flucytosine) cured (combined clinical and microbiological response) versus placebo (Amphotericin B + 5-flucytosine) and versus Mycograb + Amphotericin B alone. | day 14

SECONDARY OUTCOMES:
Safety of Mycograb versus placebo. Safety assessment will include: physical examination, vital signs, laboratory parameters, adverse events, serious adverse events. | week 10
Assess the cerebrospinal fluid (CSF) penetration of Mycograb | Days 3, 7 and 14
Determine whether Mycograb + Amphotericin B is as effective as Amphotericin B plus 5-cytosine while avoiding the potential problem of 5-cytosine toxicity. | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, South Africa, South Africa